CLINICAL TRIAL: NCT03769623
Title: A Randomized Trial of a Biolimus-Coated Balloon Versus POBA in Small Vessel Coronary Artery Disease
Acronym: Brave
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JW Medical Systems Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BIO-RISE CHINA
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Diameter: 2.0mm, 2.25mm, 2.5mm, 2.75mm Length: 10mm, 15mm, 20mm, 25mm, 30mm
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biolimus (Experimental): BA9 Drug-eluting Coronary Artery Balloon Catheter
  Interventions: Device: Biolimus
- Powerline (Active Comparator): Balloon dilated catheter
  Interventions: Device: Powerline

INTERVENTIONS:
Device: Biolimus — 103 subjects with small coronary artery disease who met the inclusion/exclusion criteria were enrolled, subjects were assigned to the treatment group of Biolimus
  Arms: Biolimus
Device: Powerline — 103 subjects with small coronary artery disease who met the inclusion/exclusion criteria were enrolled, subjects were assigned to the treatment group of Powerline
  Arms: Powerline

SUMMARY:
This study is a prospective, multicenter, randomized, blind, parallel and superiority test study. It is planned to select 206 cases of subjects with small coronary artery vessel disease who meet the inclusion/exclusion criteria. They are randomly divide them into Biolimus release coronary balloon catheter treatment group and plain old balloon angioplasty catheter (Powerline) treatment group according to the ratio of 1:1. All subjects accept clinical follow-up after operation, at 30 days, 6 months, 9 months and 12 months after operation. Follow-up with angiography is conducted at 9 months. The late lumen loss in diseased segment at 9 months after operation is the primary endpoint.

DETAILED DESCRIPTION:
The study was a prospective, multicenter, randomized, blind, parallel positive control, and superiority test study, 206 subjects with small coronary artery disease who met the inclusion/exclusion criteria were enrolled, subjects were randomly assigned to the treatment group of Biolimus and Powerline at 1:1. All subjects underwent clinical follow-up at 30 days, 6 months, 9 months, and 12 months after surgery, and angiographic follow-up at 9 months. The primary endpoint was late lumen loss at 9 months.

The study will enroll 206 subjects. The sample size determination process is as follows:

Sample size is calculated according to the primary endpoint, late lumen loss (LLL) in diseased segment at 9 months after operation. Through literature review, a Meta analysis combined 11 randomized and control study shows that the late lumen loss level of control group (POBA) in the treatment of small vessel disease is 0.54mm. Another Meta analysis shows that LLL after PTCA operation is 0.57±0.57mm. Clinical investigators and statisticians, according to literature and clinical practice, suppose that the LLL level of test group (DCB) in this study can be lowered to 0.32mm and the combined standard deviation of LLL of the two groups is estimated to be 0.50mm conservatively.

The calculation formula of sample size for parallel design and superiority test is used. In case of taking 0.025 at singles side for inspection level, taking 80% for power (1-β), and taking 0 for superiority cut-off, conduct random grouping according to the ratio of 1:1, the require sample size of each group is calculated to be 82 cases. Considering the maximum failure rate 20% in angiography follow-up (as well as the early withdrawal and random damage caused by other reasons), the planned total sample size of both groups is 206 cases finally, including 103 cases for test group (DCB) and 103 cases for control group.

ELIGIBILITY:
General inclusion criteria

1. Subjects with stable angina pectoris, unstable angina pectoris, old myocardial infarction or silent myocardial ischemia with objective evidence;
2. Subjects at the age between ≥18 and ≤75 years old;
3. Subjects without contraindications of coronary revascularization (PCI or CABG);
4. Subjects are willing to participate in the study, sign informed consent form, and accept angiography follow-up at 9 months after operation as well as clinical follow-up after operation and at 30 days, 6 months, 9 months and 12 months after operation.

Radiography inclusion criteria

1. Target lesion is primary in-situ coronary artery disease, located on 1 or 2 different coronary artery vessels, with no more than 1 target lesion on each coronary artery vessel (in case of lesion on two vessels, 2 target lesions are allowed at most);
2. Reference vessel diameter is between 2.0 mm and 2.75 mm (visual observation);
3. For non-target vessel lesion, interventional therapy needs to be conducted firstly (simultaneous therapy is required). After successful therapy, it is required to conduct random and target lesion treatment;
4. Preoperative diameter stenosis must be ≥70% or ≥50%, accompanied with corresponding ischemia of target vessel (visual observation);
5. Each target lesion of patients in test group and control group can only be treated with one trial device (Biolimus release coronary balloon catheter) or control device (Powerline balloon angioplasty catheter).

Exclusion Criteria:

General exclusion criteria

1. Any patient with myocardial infarction within one month;
2. Patients with severe congestive heart failure (NYHA Level IV severe heart failure) or severe valvular heart disease;
3. Patients with cardiogenic shock;
4. Patients with left ventricular ejection fraction of less than 35%;
5. Female patients planned for or in pregnancy (or lactation) or male patients planned for impregnation;
6. Patients with the expected lifetime of no more than 1 year or potential factors of difficulty in clinical follow-up;
7. Patients who are participating in the clinical trial of other drug or device without reaching the time limit of primary endpoint, or reaching the time limit of primary endpoint but less than 3 months;
8. Patients who plans to accept selective operation within 12 months;
9. Patients with severe liver failure (ALT and AST are larger than 3 times of the upper limit of normal value), who are judged to be not applicable to angiography by investigators;
10. Patients with severe renal failure(eGFR<30ml/minute) or such medical history, failure to comply with angiography conditions;
11. Patients with stroke, peptic ulcer or gastrointestinal bleeding within the past 6 months;
12. Patients with bleeding tendency or coagulation disorders;
13. Patients who are intolerance to aspirin and/or clopidogrel or ticagrelor or have contraindications;
14. Subjects who are intolerance or allergic to heparin, contrast agent, Biolimus, polyethylene oxide and polylactic acid - glycolic acid polymer;
15. Patients with other diseases (for instance, malignant tumor, organ grafting or candidate) or addiction history (such as alcohol, cocaine and heroin);
16. Subjects who are considered to be not applicable to be enrolled by investigators due to other reasons.

Radiography exclusion criteria

1. Evidence for extensive thrombus within target vessel;
2. Chronic total occlusion (TIMI Level 0 blood flow before operation);
3. For the left main disease and/or triple vessel disease and bypass lesion needed to be treated simultaneously, branch vessel diameter shall be ≥ 2.5mm bifurcation lesion;
4. Lesions within a distance of 3mm from circumflex branch, anterior descending branch and right coronary artery orifice;
5. After treating other vascular lesions at the same period, there are more than two lesions within the same target vessel needed to be treated;
6. There are more than 2 non-target lesions needed to be intervened or non-target lesion is not intervened before target lesion;
7. There is target vessel distortion or severe calcification lesion, so balloon catheter fails to pass it;
8. Target lesion is in-stent restenosis;
9. After predilation of target lesion, residual stenosis is ≥30% or TIMI blood flow is < Level 3, and/or there is NHBL Level C or above dissection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-04-06 (Actual)

PRIMARY OUTCOMES:
The late lumen loss | 9 months
  The late lumen loss in the lesion segment 9 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, Principal Investigator — The General Hospital of Northern Theater Command
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, Liaoning, China

REFERENCES:
- [Derived] Xu K, Fu G, Tong Q, Liu B, Han X, Zhang J, Ma G, Yang Q, Li H, Zhou Y, Jing Q, Li Y, Han Y. Biolimus-Coated Balloon in Small-Vessel Coronary Artery Disease: The BIO-RISE CHINA Study. JACC Cardiovasc Interv. 2022 Jun 27;15(12):1219-1226. doi: 10.1016/j.jcin.2022.03.024. Epub 2022 May 25. PMID 35738744